CLINICAL TRIAL: NCT01717586
Title: Pravastatin for the Prevention of Preeclampsia in High-Risk Women: A Phase I Pilot Study
Brief Title: Pravastatin for Prevention of Preeclampsia
Acronym: Statin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: University of Pittsburgh (Other); Northwestern University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-097 OPRU/OPRC Pravastatin; U54HD047891 (NIH)
Record Dates: First submitted 2012-01-03; First posted 2012-10-30 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia
Keywords: preeclampsia; pravastatin; Pravachol®; statin; high-risk pregnancy; safety; fetal morbidity and mortality; maternal morbidity and mortality; neonatal mortality; premature delivery; preemie
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth | interventions — Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pravastatin Group (Active Comparator): Pregnant women at high-risk for preeclampsia who are taking pravastatin during their pregnancy.
  Interventions: Drug: Pravastatin
- Control Group (Placebo Comparator): Pregnant women who are at high-risk for developing preeclampsia who are taking a placebo during their pregnancy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pravastatin — Comparison of different drug dosages. Women will be instructed to take a pravastatin pill everyday starting the day of randomization and ending the day of delivery. The women will be divided into three cohorts. Each cohort will receive one of the following doses of pills: 10mg or 20mg or 40mg.
  Other Names: pravastatin sodium; Brand name: Pravachol®
  Arms: Pravastatin Group
Drug: Placebo — Women will be instructed to take a placebo pill daily beginning the day of randomization and ending the day of delivery.
  Arms: Control Group

SUMMARY:
The primary purpose of this pilot study is to determine the pharmacokinetic (PK) parameters and collect preliminary safety data for pravastatin when used as a prophylactic daily treatment in pregnant women at high risk of preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia shares pathogenic similarities with adult cardiovascular diseases as well as many risk factors. Endothelial dysfunction and inflammation are fundamental for the initiation and progression of both. There is strong evidence that 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors (statins) are beneficial in primary and secondary prevention of cardiovascular mortality and other cardiovascular events. Biological plausibility as well as animal data supports a similar role for statins in preeclampsia.

Currently, there are no clinically available agents to prevent preeclampsia. However because of the below properties of statins, this class of medications could substantially contribute to preeclampsia prevention.

1. Statins pleiotropic actions on various mechanisms: reversing the angiogenic imbalance by upregulating vascular endothelial growth factor (VEGF) and placental growth factor (PlGF), and reducing the antiangiogenic factors such as soluble fms-like tyrosine kinase-1 (sFlt-1) and soluble endoglin (sEng).
2. Statins up regulation of endothelial nitric oxide synthase, leading to improved nitric oxide production in the vasculature and to activate the heme oxygenase-1/carbon monoxide (HO-1/CO) pathway, protecting the endothelium and reducing the inflammatory and oxidative insults.

The purpose of this pilot study is to evaluate the maternal-fetal safety and pharmacokinetic (PK) profiles of pravastatin when used in pregnant women at high-risk of developing preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

Documented history (review of chart or delivery note) of prior severe early onset PE in a prior pregnancy and requiring delivery ≤340/7 weeks' gestation. If in the index pregnancy, the woman was induced at the upper limit of 34 0/7 weeks of pregnancy and delivered within 48 hours in the same hospitalization, that woman could be enrolled. Women with severe PE in a pregnancy remote (greater than 2 pregnancies removed) from the current pregnancy do not qualify.

* 18 years or older with the ability to give informed consent
* Singleton pregnancy
* Normal serum transaminase (ALT and AST) concentrations in the last 6-months
* Gestational age (GA) between 12 weeks 0 days to 16 weeks 6 days based on clinical information and confirmed by an ultrasound per study procedures.
* Willingness to participate in planned PK study visits

Exclusion Criteria:

Known chromosomal, genetic, or major fetal malformations, fetal demise, or planned termination

* Patients with contraindications for statin therapy:
* Hypersensitivity to pravastatin or any component of the product
* Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes (2 x normal of serum transaminases)
* History of myopathy or rhabdomyolysis
* Patients with any of the following conditions:
* HIV positive
* Status post solid organ transplant
* Chronic renal disease/insufficiency with baseline serum creatinine ≥1.5 mg/dL
* Uterine malformations (didelphus, bicornuate, unicornate)
* Cancer
* Statin use in current pregnancy
* Current use of medications with potential drug interactions with statins, such as cyclosporine, fibrates, gemfibrozil, niacin, erythromycin, fluconazole, itraconazole, cholestyramine, digoxin, rifampin (patients will not be excluded if the drug has been discontinued, or is prescribed for a short duration of time)
* Participating in another intervention study that influences the outcomes of this study
* Plans to deliver in a non-network site

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Number and type of maternal adverse events | From the date of randomization until the date of delivery, assessed up to 210 days
  The presence of side effects and adverse events will be assessed at each study visit by:
  * a symptoms checklist
  * any other report of adverse events
  * at select visits: laboratory testing for liver function test(LFT) and creatine kinase(CK)
Number and type of fetal/neonatal adverse events | From date of birth up to discharge or 120 days after birth.
  The presence of adverse events will be assessed by evaluating
  * Fetal and neonatal death
  * Birthweight (including rate of small for gestational age)
  * Apgar scores
  * Congenital malformations
  * Auditory brainstem response (ABR) evoked potential
  * Cord blood lipid profile, AST/ALT, and CK levels
Pharmacokinetic parameters of pravastatin sodium during pregnancy | Between Pre-dose (0) and 24 hours post dose
  Timed blood and urine collection performed once between 18 wks 0 days GA and 23 wks 6 days GA and once between 30 wks 0 days GA and 33 wks 6 days GA.
  Timed blood collection intervals: pre-dose(0)and 0.5hr, 1hr, 1.5hr, 2hr, 3hr, 4hr, 6hr, 8hr post dose.
  Time urine collection intervals: pre-dose (0) and 0-4hr, 4-8hr hr post dose.
  Evaluation parameters:Maximum observed plasma concentration (Cmax) and peak time (Tmax), Steady-state area under the plasma concentration-time curve during the 24-h dosing interval (AUC0-24h), Steady-state apparent oral clearance (CL/F), Elimination half-life (t½), Renal clearance of pravastatin

CONTACTS AND LOCATIONS:
Overall Officials: Maged Costantine, MD, Principal Investigator — UTexasGalveston; Ohio State
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No
per NICHD guidelines

REFERENCES:
- [Background] Costantine MM, Cleary K, Hebert MF, Ahmed MS, Brown LM, Ren Z, Easterling TR, Haas DM, Haneline LS, Caritis SN, Venkataramanan R, West H, D'Alton M, Hankins G; Eunice Kennedy Shriver National Institute of Child Health and Human Development Obstetric-Fetal Pharmacology Research Units Network. Safety and pharmacokinetics of pravastatin used for the prevention of preeclampsia in high-risk pregnant women: a pilot randomized controlled trial. Am J Obstet Gynecol. 2016 Jun;214(6):720.e1-720.e17. doi: 10.1016/j.ajog.2015.12.038. Epub 2015 Dec 23. PMID 26723196
- [Background] Costantine MM, West H, Wisner KL, Caritis S, Clark S, Venkataramanan R, Stika CS, Rytting E, Wang X, Ahmed MS; Eunice Kennedy Shriver National Institute of Child Health and Human Development Obstetric-Fetal Pharmacology Research Centers (OPRC) Network, Bethesda, MD. A randomized pilot clinical trial of pravastatin versus placebo in pregnant patients at high risk of preeclampsia. Am J Obstet Gynecol. 2021 Dec;225(6):666.e1-666.e15. doi: 10.1016/j.ajog.2021.05.018. Epub 2021 May 24. PMID 34033812
- [Background] Costantine MM, Cleary K; Eunice Kennedy Shriver National Institute of Child Health and Human Development Obstetric--Fetal Pharmacology Research Units Network*. Pravastatin for the prevention of preeclampsia in high-risk pregnant women. Obstet Gynecol. 2013 Feb;121(2 Pt 1):349-353. doi: 10.1097/AOG.0b013e31827d8ad5. PMID 23344286
- [Derived] Costantine MM, Clifton RG, Boekhoudt TM, Lawrence K, Gyamfi-Bannerman C, Wisner KL, Grobman W, Caritis SN, Simhan HN, Hebert MF, Longo M, Saade GR; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network and the Obstetric-Fetal Pharmacology Research Centers Network. Long-term neurodevelopmental follow-up of children exposed to pravastatin in utero. Am J Obstet Gynecol. 2023 Aug;229(2):153.e1-153.e12. doi: 10.1016/j.ajog.2023.02.016. Epub 2023 Feb 24. PMID 36842489